CLINICAL TRIAL: NCT07089836
Title: ALPCO Syphilis-T and Syphilis-NT CLIA Kits: Detection of Antibodies to Treponema Pallidum and Against Lipoidal Antigens in Human Serum and Plasma
Brief Title: This Study Evaluates the ALPCO Syphilis-T and Syphilis-NT CLIA Kits for Detecting Syphilis Antibodies in Serum and Plasma. Samples From At-risk, HIV-positive, Pregnant, and Healthy Individuals Will Assess Assay Performance Versus Established Comparator Tests.
Status: Recruiting | Type: Observational
Sponsor: American Laboratory Products Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CPSP-2025-020
Record Dates: First submitted 2025-07-22; First posted 2025-07-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Treponema Pallidum; Treponema Pallidum Infection; Syphilis Infection; Serum; Plasma; Blooddraw; Sexually Transmitted Infection (STI)
Keywords: Non Treponema; Treponema; Syphilis; Sample Collection; Treponema pallidum; Non-treponemal test; Chemiluminescent immunoassay; HIV-positive; Pregnant women; Blood sample collection
MeSH Terms: conditions — Treponemal Infections; Syphilis; Sexually Transmitted Diseases; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples will be collected from participants via venipuncture. These samples will be used to evaluate the performance of the investigational syphilis diagnostic assays. Retained biospecimens will not be used for DNA extraction and will be stored under appropriate conditions for future diagnostic validation studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Syphilis-Positive Patients: Individuals with a current or prior diagnosis of syphilis.
  Interventions: Device: ALPCO Syphilis-T; Device: ALPCO Syphilis-NT CLIA Kits
- HIV-Positive Patients: Individuals diagnosed with HIV (may or may not overlap with other cohorts).
  Interventions: Device: ALPCO Syphilis-T; Device: ALPCO Syphilis-NT CLIA Kits
- Pregnant Individuals: Pregnant participants across all trimesters.
  Interventions: Device: ALPCO Syphilis-T; Device: ALPCO Syphilis-NT CLIA Kits
- Apparently Healthy Individuals: Participants with no known history or symptoms of syphilis.
  Interventions: Device: ALPCO Syphilis-T; Device: ALPCO Syphilis-NT CLIA Kits

INTERVENTIONS:
Device: ALPCO Syphilis-T — Detection of antibodies to Treponema pallidum in human serum and plasma
Device: ALPCO Syphilis-NT CLIA Kits — Detection of antibodies to lipoidal antigens in human serum and plasma

SUMMARY:
This study will evaluate the clinical performance of two investigational diagnostic kits developed by ALPCO: the Syphilis-T CLIA Kit and the Syphilis-NT CLIA Kit. These kits are designed to detect antibodies to Treponema pallidum and non-treponemal lipoidal antigens, respectively, in human serum and plasma using the automated KleeYa platform. The study will collect and analyze blood samples from individuals suspected of having syphilis, those at high risk, HIV-positive patients, pregnant individuals, and healthy controls. The aim is to determine the kits' Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA) compared to established reference assays.

DETAILED DESCRIPTION:
This is a multicenter, prospective clinical collection study designed to evaluate the diagnostic performance of the ALPCO Syphilis-T and Syphilis-NT CLIA Kits. The study will enroll individuals undergoing routine syphilis testing, those with a history of syphilis, HIV-positive individuals, pregnant individuals, and healthy volunteers. Blood samples will be collected, processed, and tested across up to three clinical sites using the investigational kits. Reference results will be determined using validated, FDA-cleared treponemal and non-treponemal tests. For the treponemal assay, results will be considered accurate if they match at least two of the three reference tests. The primary objective is to demonstrate that both kits meet or exceed prespecified performance criteria, including ≥95% positive and negative percent agreement (≥99% NPA for the non-treponemal kit), with the lower bound of the 95% confidence interval at or above 90%.

ELIGIBILITY:
Inclusion Criteria:

* Male, Female, or Other(s)
* Patients undergoing routine syphilis testing (asymptomatic at risk, suspected with symptoms, prior history of syphilis, high risk for syphilis) or previously diagnosed with syphilis through a test performed in an accredited laboratory.
* Participants must be willing to provide the required blood samples for the clinical study, in addition to any samples requested by their physician.
* Pregnant individuals and children (under 22): 1 clinical study tube of blood.
* All other participants (excluding pregnant individuals and children): 2 clinical study tubes of blood.
* Participants must be able and willing to sign the informed consent form (ICF).
* Participants aged 13 to 17 will be asked to sign an assent form. Written parental or guardian consent will also be required prior to enrollment. The assent form will use age-appropriate language and be reviewed with the participant before any procedures.

Exclusion Criteria:

* Patients currently being treated with antibiotics or completed a course of antibiotics within the past 30 days
* Patients with pre-existing conditions that would make blood collection difficult or harmful
* If the samples are not collected in strict accordance with the established sampling protocol, as determined by the study team.
* Any medical, psychological, or social condition that, in the judgment of the investigator, could interfere with the participant's ability to comply with study requirements, or pose a risk to their safety, or compromise the integrity of the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of syphilis, at high-risk for syphilis, or scheduled for routine syphilis related serological testing will be enrolled in the clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Percent Agreement of the ALPCO Syphilis-T and Syphilis-NT CLIA Kits | 6 months
  Evaluate the clinical performance of the ALPCO Syphilis-T and Syphilis-NT CLIA Kits in detecting antibodies to Treponema pallidum and lipoidal antigens, by comparing results against established comparator assays. Success is defined as meeting or exceeding pre-specified thresholds for Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA), with lower bounds of the 95% confidence interval ≥90%.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Chemidox Clinical Trials California, Lancaster, California
  - Folio Clinical Research, Los Angeles, California
  - Segel Trials, North Miami, Florida
  - IMA Clinical Research - St.Petersburg, St. Petersburg, Florida
  - Chemidox Tx LLC, Houston, Texas
  - VAST Clinical Research, Mesquite, Texas

IPD SHARING:
Plan to Share IPD: No